CLINICAL TRIAL: NCT01257503
Title: Randomized Controlled Trial of a Homeopathic Cold Remedy for Children
Brief Title: Homeopathic Cold Remedy for Children Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Standard Homeopathic Company (Industry)
Responsible Party: Principal Investigator, James Taylor, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 39489-D
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2015-01-02 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2014-12

CONDITIONS: Upper Respiratory Tract Infections
Keywords: children; upper respiratory tract infections; homeopathy
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homeopathic cold remedy (Experimental): 5 ml of homeopathic cold remedy given by mouth up to 6 times per day as needed for cold symptoms
  Interventions: Drug: Hyland's Cold 'n Cough 4 kids
- placebo (Placebo Comparator): 5 ml of placebo given by mouth up to 6 times per day as needed for cold symptoms
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Hyland's Cold 'n Cough 4 kids — 5 ml PO q4h prn cold symptoms
  Arms: Homeopathic cold remedy
Drug: placebo — liquid made to look like the active homeopathic remedy
  Arms: placebo

SUMMARY:
A randomized controlled trial of a commercially available homeopathic cold remedy will be conducted. A total of 400 children, 2-5 years old, diagnosed with an upper respiratory tract infection will be randomized to receive either the homeopathic remedy or placebo. Parents of study children will administer 5 ml of the study medication up to 6 times per day as needed to treat cold symptoms. One hour after giving a dose the parent will rate change in symptoms (for up to the first 10 doses). In addition, parents will rate their child's overall symptom severity and functional status over the first 3 days of the cold. It is postulated that children receiving the active homeopathic remedy will have better symptom relief and that their symptom severity and functional status will improve more rapidly than those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of upper respiratory tract infection
* duration of symptoms < 7 days
* Parent who speaks English

Exclusion Criteria:

* history of asthma
* on any prescribed medication
* prescribed any medication other than acetaminophen or ibuprofen at index visit
* use of homeopathic remedy within 48 hours of index visit

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 263 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center- Roosevelt Pediatric Care Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Homeopathic Cold Remedy | Placebo
Started | 133 | 130
Returned Symptom Diaries | 80 | 83
Returned Dosage Logbooks | 75 | 80
Completed | 125 (Completed defined as participants who completed telephone follow-up at end of study period) | 119 (Completed defined as participants who completed telephone follow-up at end of study period)
Not Completed | 8 | 11
Not completed — Lost to Follow-up | 7 | 10
Not completed — Over 5 years old at enrollment | 0 | 1
Not completed — strep culture positive at enrollment | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients enrolled. Age data were analyzed on 127 participants in the placebo group since exact data were missing for 2 participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Homeopathic Cold Remedy | Placebo | Total
Number analyzed (Participants) | 132 | 129 | 261
Age, Categorical [Count of Participants; unit: Participants] — exact age information missing on 2 participants in placebo group, noted to be 2-5 years old
  Participants
    <=18 years | 132 | 129 | 261
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (1.1) | 3.5 (1.1) | 3.5 (1.1)
Gender [Number; unit: participants] — Gender information missing on 1 participant randomized to the homeopathic cold remedy group
  participants
    Female | 64 | 62 | 126
    Male | 67 | 67 | 134
Region of Enrollment [Number; unit: participants]
  United States | 132 | 129 | 261
baseline cold symptom score [Mean (Standard Deviation); unit: units on a scale] — sum of scores for runny nose severity, sneeze severity, cough severity and congestion severity rated by parent at study entry. For each symptom, possible scores range from 0 to 3, with 3 indicating most severe. Baseline cold score missing on 1 participant in the homeopathic cold remedy group
  units on a scale | 5.4 (1.8) | 5.2 (1.8) | 5.3 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Cold Symptoms
Description: Parents measured change in runny nose, cough, nasal congestion and sneezing severity one hour after administering a dose of study medication up to the first 10 doses of study medication. Change in symptom rated from 0 to 6, with 0 indicative of the symptom being much worse and 6 indicative of the symptom being much improved. The unit of analysis for each outcome was doses of medication. Each participant could contribute data on 0 - 10 doses.
Time Frame: Parents assessed change in symptom 1 hour after a dose of study medication
Population: Data are from logbooks returned by participants. For each participant, data on response to up to 10 doses were collected. Not every symptom was present at each dose. Change in runny nose assessed after 819 doses, sneeze 456 doses, cough 772 doses, congestion 845. For category title, first n= homeopathic cold remedy, second n= placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: doses
Arm/Group | Homeopathic Cold Remedy | Placebo
Number analyzed (Participants) | 75 | 80
Number analyzed (doses) | 502 | 480
units on a scale
  runny nose (n=433, 386) | 3.7 (1.3) | 3.7 (1.0)
  sneeze (n=219, 237) | 3.9 (1.2) | 3.9 (1.2)
  cough (n=399, 373) | 3.8 (1.2) | 3.8 (1.2)
  congestion (n=409, 436) | 3.8 (1.1) | 3.7 (1.0)
Statistical Analysis 1: Comparison: Homeopathic Cold Remedy vs Placebo; change in runny nose; Test type: Superiority or Other; p = .86, Regression, Linear; generalized estimating equations used to account for multiple doses in same participant
Statistical Analysis 2: Comparison: Homeopathic Cold Remedy vs Placebo; change in sneeze; Test type: Superiority or Other; p = .89, Regression, Linear; generalized estimating equations used to account for multiple doses in single participant
Statistical Analysis 3: Comparison: Homeopathic Cold Remedy vs Placebo; change in cough; Test type: Superiority or Other; p = .45, Regression, Linear; generalized estimating equations used to account for multiple doses in single participant
Statistical Analysis 4: Comparison: Homeopathic Cold Remedy vs Placebo; change in congestion; Test type: Superiority or Other; p = .82, Regression, Linear; generalized estimating equations used to account for multiple doses in single participant

2. Secondary Outcome: Change in Non-specific Symptoms
Description: Parents measured change in severity of irritability, lethargy, fussiness, and appetite one hour after administering a dose of study medication up to the first 10 doses of study medication. Change in symptom rated from 0 to 6, with 0 indicative of the symptom being much worse and 6 indicative of the symptom being much improved. The unit of analysis for each outcome was doses of medication. Each participant could contribute data on 0 - 10 doses.
Time Frame: Parents assessed change in symptom 1 hour after dose of study medication
Population: Data are from logbooks returned by participants. For each participant, data on response to up to 10 doses were collected. Not every symptom was present at each dose. Change in irritability assessed after 510 doses, lethargy 414, fussiness 501, appetite 618. For category title, first n= homeopathic cold remedy, second n= placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: doses
Arm/Group | Homeopathic Cold Remedy | Placebo
Number analyzed (Participants) | 75 | 80
Number analyzed (doses) | 502 | 480
units on a scale
  irritability (n= 272, 238) | 3.6 (1.1) | 3.5 (1.2)
  lethargy (n=213, 201) | 3.6 (1.1) | 3.6 (1.1)
  fussiness (n=262, 239) | 3.6 (1.2) | 3.5 (1.2)
  appetite (n=312, 306) | 3.6 (1.0) | 3.5 (1.1)
Statistical Analysis 1: Comparison: Homeopathic Cold Remedy vs Placebo; change in irritability; Test type: Superiority or Other; p = .61, Regression, Linear; Generalized estimating equations used to account for multiple doses in single participant
Statistical Analysis 2: Comparison: Homeopathic Cold Remedy vs Placebo; change in lethargy; Test type: Superiority or Other; p = .97, Regression, Linear; Generalized estimating equations used to account for multiple doses in single participant
Statistical Analysis 3: Comparison: Homeopathic Cold Remedy vs Placebo; change in fussiness; Test type: Superiority or Other; p = .79, Regression, Linear; Generalized estimating equations used to account for multiple doses in single participant
Statistical Analysis 4: Comparison: Homeopathic Cold Remedy vs Placebo; change in appetite; Test type: Superiority or Other; p = .81, Regression, Linear; Generalized estimating equations used to account for multiple doses in single participant

3. Secondary Outcome: Functional Status
Description: Change in functional status of child during the 7-10 days after the index visit for an upper respiratory tract infection. Parents rated 5 activities (vigorous activity, activities that require concentration, activities with family or friends, appetite and sleep) daily for 3 days in their child and again at the 7-10 day follow-up. Functional status scores range from 0 to 15, with higher scores indicative of better functional status.
Time Frame: 10 days
Population: Participants who completed follow-up and had valid data for functional outcome. Data on functional status analyzed on days 1-3 for participants who returned symptom diaries including 145 on day 1, 142 on day 2 and 130 on day 3. For category title, first n= homeopathic cold remedy, second n= placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Homeopathic Cold Remedy | Placebo
Number analyzed (Participants) | 123 | 117
units on a scale
  functional status day 1 (n=68, 77) | 11.0 (3.5) | 10.4 (3.1)
  functional status day 2 (n=72, 70) | 11.7 (3.4) | 11.8 (3.4)
  functional status day 3 (n= 62, 68) | 12.7 (3.0) | 12.5 (3.0)
  functional status at follow-up (n=123, 117) | 14.2 (1.7) | 13.7 (2.7)
Statistical Analysis 1: Comparison: Homeopathic Cold Remedy vs Placebo; functional status day 1; Test type: Superiority or Other; p = .16, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Homeopathic Cold Remedy vs Placebo; functional status day 2; Test type: Superiority or Other; p = .70, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Homeopathic Cold Remedy vs Placebo; functional status day 3; Test type: Superiority or Other; p = .77, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Homeopathic Cold Remedy vs Placebo; functional status at 7-10 day follow-up; Test type: Superiority or Other; p = .41, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Health Status
Description: Change in health status of child during the 7-10 days after the index visit for an upper respiratory tract infection. Parents rated health status on 1-10 scale with 1 indicating perfect health and 10 indicating very sick. Health status rated on first 3 days of study and again at the 7-10 day follow-up
Time Frame: 10 days
Population: Health status on those with follow-up data and a valid score for health status. Health status also assessed in participants who returned symptom diaries including 152 on day 1, 142 on day 2 and 132 on day 3. For category title, first n= homeopathic cold remedy, second n= placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Homeopathic Cold Remedy | Placebo
Number analyzed (Participants) | 125 | 117
units on a scale
  health status day 1 (n=75, 77) | 4.4 (1.9) | 4.9 (2.0)
  health status day 2 (n=72,70) | 3.8 (1.9) | 4.1 (1.8)
  health status day 3 (n=63, 69) | 3.2 (2.0) | 3.4 (1.7)
  health status at follow-up (n=125, 117) | 2.5 (1.7) | 2.5 (1.6)
Statistical Analysis 1: Comparison: Homeopathic Cold Remedy vs Placebo; health status day 1; Test type: Superiority or Other; p = .10, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Homeopathic Cold Remedy vs Placebo; health status day 2; Test type: Superiority or Other; p = .28, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Homeopathic Cold Remedy vs Placebo; health status day 3; Test type: Superiority or Other; p = .26, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Homeopathic Cold Remedy vs Placebo; health status at follow-up; Test type: Superiority or Other; p = .88, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Overall Symptom Severity
Description: Change in cold symptoms of child during the 7-10 days after the index visit for an upper respiratory tract infection. Parents assessed severity of runny nose, cough, sneeze and congestion in their child using a 0-3 scale for each symptom, 0=none to 3= severe. Cold score is sum of scores for each symptom. Parents assessed cold score twice daily on study days 1-3 and at the 7-10 day follow-up
Time Frame: 10 days
Population: Data analyzed on participant who completed 7-10 day follow-up and had valid cold scores. Data also analyzed twice daily on those participants who returned symptom diaries including: day 1 (153, 148), day 2 (146,138), and day 3 (136, 126). For category title, first n= homeopathic cold remedy, second n= placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Homeopathic Cold Remedy | Placebo
Number analyzed (Participants) | 123 | 117
units on a scale
  day 1 assessment 1 (n=73, 80) | 4.6 (2.2) | 5.5 (2.3)
  day 1 assessment 2 (n=72, 76) | 4.2 (2.4) | 5.0 (2.0)
  day 2 assessment 1 (n=73, 73) | 3.7 (2.2) | 4.0 (2.0)
  day 2 assessment 2 (n=69, 69) | 3.4 (2.3) | 4.0 (2.2)
  day 3 assessment 1 (n=68, 68) | 3.0 (2.5) | 3.0 (2.3)
  day 3 assessment 2 (n= 60, 66) | 2.8 (2.5) | 3.0 (2.3)
  follow-up (n= 123, 117) | 2.4 (2.6) | 2.0 (2.0)
Statistical Analysis 1: Comparison: Homeopathic Cold Remedy vs Placebo; cold score day 1 assessment 1; Test type: Superiority or Other; p = .02, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Homeopathic Cold Remedy vs Placebo; cold score day 1 assessment 2; Test type: Superiority or Other; p = .01, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Homeopathic Cold Remedy vs Placebo; day 2 assessment 1; Test type: Superiority or Other; p = .25, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Homeopathic Cold Remedy vs Placebo; cold score day 2 assessment 2; Test type: Superiority or Other; p = .15, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Homeopathic Cold Remedy vs Placebo; cold score day 3 assessment 1; Test type: Superiority or Other; p = .88, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Homeopathic Cold Remedy vs Placebo; cold score day 3 assessment 2; Test type: Superiority or Other; p = .35, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Homeopathic Cold Remedy vs Placebo; cold score at 7-10 day follow-up; Test type: Superiority or Other; p = .36, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Data were collected during the study period and at the follow-up phone call scheduled 7-10 days after enrollment
Description: Parents were asked to record any side effects after each dose of study medications. Parents also asked about side effects during follow-up phone call.
Arm/Group | Homeopathic Cold Remedy | Placebo
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/130
Other Adverse Events (participants affected / at risk) | 0/133 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days